CLINICAL TRIAL: NCT07188753
Title: OLDEP-TBS - Randomized Controlled Trial Testing the Efficacy of Transcranial Magnetic Stimulation by Accelerated & High-dose Theta-burst, Functional Imaging Guided, in the Treatment of Depression in Elderly Subjects With Cognitive Impairment
Brief Title: Randomized Controlled Trial Testing the Efficacy of Transcranial Magnetic Stimulation by Accelerated & High-dose Theta-burst, Functional Imaging Guided, in the Treatment of Depression in Elderly Subjects With Cognitive Impairment
Acronym: OLDEP-TBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35RC22_9819_OLDEP-TBS
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Treatment Resistant Depression; Elderly Depression (≥65y.o.)
Keywords: transcranial magentic stimulation; personalized targeting; depression; elderly; old-age depression; treatment resistant; accelerated TMS; iTBS; theta birst stimulation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (participant, operator, investigator) Randomisation code sent to the administrator administering the treatment. Cool 865 Active/Placebo coil
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): active transcranial magnetic stimulation using accelerated (aiTBS)
  Interventions: Other: transcranial magnetic stimulation by accelerated & high-dose theta-burst, functional imaging guided, i
- Control group (Placebo Comparator): Placebo transcranial magnetic stimulation (Sham stimulation)
  Interventions: Other: transcranial magnetic stimulation by accelerated & high-dose theta-burst, functional imaging guided, i

INTERVENTIONS:
Other: transcranial magnetic stimulation by accelerated & high-dose theta-burst, functional imaging guided, i — Participants will then be treated with 1,800 pulses of iTBS (3-pulse 50-Hz bursts at 5-Hz for 2-second trains, with trains every 10 seconds) per session at 90% resting motor threshold and depth-adjustment to the personalized functional target. Each session will last 10 min followed by a 50-minute intersession interval. Ten sessions will be applied per day (18,000 pulses/day) for 5 consecutive days (90,000 total pulses).

SUMMARY:
This trial aims at testing a new intensive, personalized functional targeting, transcranial magnetic stimulation technique for elderly patients (aged ≥ 65 years) suffering from a current treatment resistant depressive episode to at least one antidepressant, and suffering from significant secondary cognitive impairment.

The intervention will be based on an accelerated neuromodulation technique using intermittent theta bursts (aiTBS) guided by a personalised funcitonal target within the left dorsolateral prefrontal cortex (DLPFC), using the SAINT® technology, which was recently cleared by the FDA.

DETAILED DESCRIPTION:
Depression in older adults is often associated with cognitive impairment. Executive dysfunction exposes patients to poor response to antidepressants, increased risk of relapse and suicide, and greater disability. Depression doubles the risk of developing dementia in later life.

Late-onset depression is considered more difficult to treat due to low tolerance to standard antidepressant treatments, which prevents dose optimisation. Late-onset depression is considered more difficult to treat due to poor tolerance to standard antidepressant treatments, which prevents dose optimisation.

Furthermore, antidepressants are not optimal for improving cognitive function. Thus, antidepressant therapies are limited in terms of efficacy or tolerance, leading to persistent depressive symptoms and cognitive deficits that impact daily functioning, quality of life, and even independence.

Transcranial magnetic stimulation, a focused non-pharmacological antidepressant therapy, is a promising alternative. Several meta-analyses have demonstrated its efficacy as an antidepressant treatment and its potential for treating mild cognitive impairment. However, these studies have encountered certain limitations, such as small sample sizes and heterogeneity. Recently, a randomised controlled trial testing an accelerated form of intermittent theta burst stimulation (aiTBS) in adults with treatment-resistant depression demonstrated a high remission rate of approximately 80% (with effect sizes ranging from [1.4-1.8]). This technique has a good tolerance profile.

Overall, aiTBS treatment has several potentially beneficial aspects for depression in older adults: efficacy, rapid onset of action, and good tolerability. Such a technique could prevent the negative impact of depression and cognitive impairment on the quality of life and independence of older adults with depression.

In this randomised controlled trial (RCT), the investigators aim to test the efficacy of aiTBS treatment guided by functional connectivity at rest in elderly patients suffering from major depressive disorder (MDD) in a major depressive episode (MDE) and cognitive impairment. The investigators hypothesise that active aiTBS treatment will be superior to placebo aiTBS treatment in improving depressive and cognitive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, of ages ≥ 65 years at the time of screening
2. Currently diagnosed with either Major Depressive Disorder (MDD) and meets criteria for a current Major Depressive Episode (MDE) according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5).
3. Patients that don't meet the treatment response criteria according to antidepressant treatment history form (ATHF) for whom a switch to another ATD is required.
4. rTMS/iTBS naïve.
5. Access to ongoing psychiatric care before and after completion of the study.
6. Access to clinical rTMS after completion of the study.
7. In good general health, as evidenced by medical history (i.e. any ongoing serious and vital medical condition).
8. Having signed a free, informed and written consent
9. Patients that have a valid health insurance and are affiliated to or beneficiary of a social security system.
10. Montgomery and Asberg Depression Rating Scale (MADRS) score of ≥ 20 at screening.
11. MoCA total score ≤ 26.
12. Comply with eligibility criteria checklist (Appendix 3)

Exclusion Criteria:

1. Major cognitive disorder according to DSM-5 criteria.
2. The presence or diagnosis of prominent (primary) anxiety disorder, personality disorder, or dysthymia.
3. Bipolar Affective Disorder I & II and primary psychotic disorders.
4. Autism Spectrum disorder or Intellectual Disability.
5. A diagnosis of obsessive-compulsive disorder (OCD).
6. Current moderate or severe substance use disorder (according to DSM-5 criteria) or demonstrating signs of acute substance withdrawal.
7. Any history of ECT (greater than 8 sessions) without meeting response criteria.
8. No recent (during the current depressive episode) or concurrent use of a rapid acting antidepressant agent (i.e., ketamine or a course of ECT).
9. History of significant neurologic disease, including Parkinson's or Huntington's disease, brain tumor, unexpected seizure/epilepsy disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma (having caused a coma and/or requiring specific hospital care, and/or with abnormal brain imaging).
10. Untreated or insufficiently treated dysthyroidism (TSH range 0.4-4mUI/l).
11. Treatment with another investigational drug or other intervention within the study period.
12. Any other condition deemed by the PI to interfere with the study or increase risk to the participant.
13. Contraindications to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion).
14. Contraindications to Magnetic Resonance Imaging (MRI) (ferromagnetic metal in their body).
15. Participants taking certain psychoactive medications will be assessed for safety by the PI, due to potential for increase of seizure risk (e.g., clozapine) and change in cortical excitability (e.g. anticonvulsant, benzodiazepines). A maximum daily dose of 2mg lorazepam equivalent will be accepted.
16. Persons referred in articles L.1121-5 to L.1121-8 and L.1122-2 of the Public Health Code: Pregnant women, women in labour and breastfeeding mothers Person deprived of liberty for judicial or administrative decision, adult person under legal protection (any form of public guardianship).
17. Mini Mental Status Examination (MMSE) score < 21.
18. Current severe insomnia (must sleep a minimum of 5 hours each night before stimulation).
19. Current mania or psychosis.
20. Endorses clinically significant explicit suicidal cognitions (score ≥ 6 on the Beck Suicide Scale [BSS] self-report).
21. Any current substance abuse that is clinically elicited or based on urine/breathalyzer screening deemed by the PI to be critical from a safety standpoint.
22. Depth-adjusted aiTBS treatment dose > 65% maximum stimulator output (MSO).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2031-06-15 (Estimated); Study Completion 2031-12-15 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of aiTBS, as compared to sham stimulation, on depressive symptoms at one-month visit (35+/-3 days after the last day of treatment). | at one-month visit (35+/-3 days after the last day of treatment)
  Montgomery and Asberg Depression Rating Scale (MADRS) (min:0 / max:60)

SECONDARY OUTCOMES:
To determine the effect of aiTBS, as compared to sham stimulation on depressive symptoms at two-month post-intervention | at two-month post-intervention (F+65D (+/-3D) after the last day of treatment).
  Montgomery and Asberg Depression Rating Scale (MADRS) (min:0 / max:60)
To determine the effect of aiTBS, as compared to sham stimulation | at six-month post-intervention (F+180D(+/-6D) after the last day of treatment)
  Montgomery and Asberg Depression Rating Scale (MADRS) (min:0 / max:60)
To determine the effect of aiTBS, as compared to sham stimulation | at one month post-intervention (+35D (+/-3D) after the last day of treatment).
  MATTIS (global cognitive functioning) score
To determine the effect of aiTBS, as compared to sham stimulation | at two-month post-intervention (F+65D (+/-3D) after the last day of treatment)
  MATTIS (global cognitive functioning) score
To determine the effect of aiTBS, as compared to sham stimulation on global cognitive functioning, at six-month post-intervention visit. | at six-month post-intervention(F+180D(+/-6D) after the last day of treatment)
  MATTIS (global cognitive functioning) score

OTHER OUTCOMES:
To determine the effect of aiTBS, as compared to sham stimulation on depressive symptoms at immediate post visit | at immediate post visit (3 or 4 Day after the last day of treatment)
  Montgomery and Asberg Depression Rating Scale (MADRS) (min:0 / max:60)
To determine the effect of aiTBS, as compared to sham stimulation on factors associated with treatment resistance at immediate, one-month, two-month, and six-month post-intervention in depression and suicide risk - such as anhedonia | at immediate, one-month, two-month, and six-month post-intervention
  SHAPS - clinician rated (anhedonia scale) score (min:0 / max:14)
To determine the effect of aiTBS, as compared to sham stimulation on factors associated with treatment resistance at immediate, one-month, two-month, and six-month post-intervention in mental pain, loneliness | at immediate, one-month, two-month, and six-month post-intervention
  Visual Analogic Scale for Mental Pain (VAS-MP) (min: 0 =smallest possible - max:10 = largest possible)
To determine the effect of aiTBS, as compared to sham stimulation on factors associated with treatment resistance at immediate, one-month, two-month, and six-month post-intervention in oneliness | at immediate, one-month, two-month, and six-month post-intervention
  BHS (hopelessness) (min:0 / max:20)
To determine the effect of aiTBS, as compared to sham stimulation on quality of life | at two-month, and six-month post-intervention visit
  SF - 36 (quality of life)
To determine the effect of aiTBS, as compared to sham stimulation on autonomy at two-month, and six-month post-intervention visit | at two-month, and six-month post-intervention visit
  Independent Living Scale (ILS) (Tremblay et al., 2021) (min:0 / max:140)
To determine the moderating effect of treatment resistance severity on the antidepressant effect of aiTBS at two-month post visit. | at two-month post visit.
  The treatment severity will be measured by the Maudsley Staging Model (min =0 ; max =15)
To monitor any medication change that may occur during the follow-up period (at immediate, one-month, two-month, and six-month post-intervention). | at immediate, one-month, two-month, and six-month post-intervention)
  Medication change (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie BATAIL, M.D.,Ph.D., Principal Investigator — C. H. GUILLAUME REGNIER RENNES; Bruno MILLET, PH-PD, Principal Investigator — APHP- LA PITIE; Ghina HARIKA GERMANEAU, MD, Principal Investigator — Centre Hospitalier Henri Laborit; Maud ROTHARMEL, MD, Principal Investigator — CHS DU ROUVRAY SOTTEVILLE-LES-ROUEN; Samuel BULTEAU, MD, Principal Investigator — Nantes University Hospital; Noomane BOUAZIZ, MD, Principal Investigator — EPS VILLE EVRARD; Moussa CHALAH, MD, Principal Investigator — GHU PARIS; David SZEKELY, MD, Principal Investigator — Centre Hospitalier Princesse Grace